CLINICAL TRIAL: NCT00086723
Title: Phase I/II Trial of In Vivo Angiostatin Generation With Tissue Plasminogen Activator (tPA) and Captopril in Patients With Progressive, Metastatic Cancer
Brief Title: In Vivo Angiostatin Generation Using Tissue Plasminogen Activator and Captopril in Treating Patients With Progressive Metastatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NCI 00B9; NU-NCI-00B9
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Tissue Plasminogen Activator; Captopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: recombinant tissue plasminogen activator
Drug: captopril

SUMMARY:
RATIONALE: Tissue plasminogen activator and captopril may help the body generate angiostatin. Angiostatin may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: This phase I/II trial is studying the side effects and best dose of tissue plasminogen activator and captopril and to see how well they work in treating patients with progressive metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and toxicity of captopril and tissue plasminogen activator (tPA) in patients with progressive metastatic cancer.
* Determine the in vivo generation of angiostatin by western analysis in patients treated with this regimen.

Secondary

* Determine the antitumor effect of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive tissue plasminogen activator (tPA) IV over 6 hours and oral captopril twice daily on days 1-5. Courses repeat every 14 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 2 additional courses beyond CR.

Cohorts of 3-6 patients receive escalating doses of tPA and captopril until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Not specified.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of progressive metastatic cancer, excluding hematologic malignancies (i.e., leukemia or lymphoma)
* Measurable disease not required
* Must have received at least 1 prior systemic treatment for metastatic disease
* No known CNS involvement

  * CNS involvement allowed provided it is successfully controlled by prior surgery or radiotherapy and there is no current requirement for corticosteroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding diathesis

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 3 times upper limit of normal
* Albumin normal
* PT and aPTT normal
* Fibrinogen > lower limit of normal

Renal

* Creatinine no greater than 1.8 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No history of stroke, transient ischemic attack, or symptoms of cerebral ischemia
* No history of angioedema with captopril
* No severe or uncontrolled hypertension (i.e., systolic blood pressure greater than 180 mm Hg or diastolic blood pressure greater than 110 mm Hg)
* No congestive heart failure requiring therapy
* No chronic hypotension (e.g., systolic blood pressure less than 100 mm Hg)

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* Potassium no greater than 5.2 mmol/L
* No active internal bleeding
* No history of seizures
* No psychiatric disorder that would preclude the giving of informed consent or study follow-up
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled or active bacterial, viral, or invasive fungal infection
* No recent trauma
* No medical indication for anticoagulation
* No contraindication to captopril

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior biologic therapy
* No concurrent immunomodulator therapy

Chemotherapy

* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior endocrine therapy

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery

* See Disease Characteristics
* No recent intracranial or intraspinal surgery
* No concurrent surgery

Other

* More than 48 hours since prior anticoagulation agents (e.g., warfarin or heparin)
* More than 3 weeks since prior investigational agents
* No concurrent anticoagulation agents, aspirin, or nonsteroidal anti-inflammatory drugs
* No other concurrent investigational agent
* No concurrent phenytoin, phenobarbital, or other antiepileptic prophylaxis
* Concurrent bisphosphonates allowed for metastatic bone disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Angiostatin production

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States